CLINICAL TRIAL: NCT00574756
Title: The Effect of Ranolazine on Echocardiographic Indices of Diastolic Dysfunction
Brief Title: Effect of Ranolazine on Echocardiographic Indices of Diastolic Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070480
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Ranolazine; Diastolic Heart Failure; Tissue Doppler Ultrasound; Echocardiography
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Other): Active drug for 2 weeks, then washout period for 2 weeks, then placebo for 2 weeks
  Interventions: Drug: ranolazine
- 2 (Other): Placebo for 2 weeks, then washout for 2 weeks, then ranolazine for 2 weeks
  Interventions: Drug: ranolazine

INTERVENTIONS:
Drug: ranolazine — extended release 500 mg twice a day for two weeks
  Other Names: Ranexa

SUMMARY:
The purpose of this study is to evaluate the effects of ranolazine, an FDA-approved medication for the treatment of angina, on heart function by using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Moderate of severe diastolic dysfunction, E/Ea>12
* Preserved systolic function
* NYHA Class I-II

Exclusion Criteria:

* QTc >450 msec at enrollment
* Taking medications that prolong QT interval or are potent inhibitors of CYP3A
* Significant coronary artery disease
* Severe valvular disease
* Hepatic disease
* Severe kidney disease
* Women of childbearing age
* Prior serious ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in E/Ea | 2 weeks

SECONDARY OUTCOMES:
changes in mitral inflow parameters (E, A, IVRT, DT) | 2 weeks
Changes in tissue doppler parameters (Ea, Aa) | 2 weeks
Changes in pulmonary venous inflow (S, D, a reversal) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DeMaria, MD, Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD Medical Center, San Diego, California, United States